CLINICAL TRIAL: NCT00005967
Title: A Dose Finding Study of R115777 (NSC 702818) in Patients With Advanced Hematologic Malignancies
Brief Title: Tipifarnib in Treating Patients With Advanced Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02342; UCCRC-10294; NCI-42; CDR0000067950 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2004-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; polycythemia vera; primary myelofibrosis; essential thrombocythemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Lymphoma, B-Cell, Marginal Zone | interventions — tipifarnib

ARMS (1):
- Arm I (Experimental): Patients receive oral tipifarnib twice daily for 21 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 1 course of therapy, patients may receive subsequent therapy at the maximum tolerated dose at the investigator's discretion.
  Interventions: Drug: tipifarnib

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
Randomized phase I trial to study the effectiveness of tipifarnib in treating patients who have advanced hematologic cancer. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the relationship between tipifarnib dose and inhibition of farnesylation in malignant cells of patients with advanced hematologic malignancies.

II. Determine the safety profile of this drug in this patient population. III. Determine the clinical activity of this drug in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 4 dose levels.

Patients receive oral tipifarnib twice daily for 21 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 1 course of therapy, patients may receive subsequent therapy at the maximum tolerated dose at the investigator's discretion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hematologic malignancy refractory to standard therapy or for which no known effective therapy exists

  * Hodgkin's or non-Hodgkin's lymphoma

    * Known bone marrow involvement
  * Acute myeloid leukemia
  * Chronic myelogenous leukemia

    * Chronic phase

      * No significant symptoms after treatment
      * No features of accelerated phase or blastic phase
    * Accelerated phase

      * WBC difficult to control with conventional busulfan or hydroxyurea in terms of dose requirement or shortening of intervals between courses
      * Rapid doubling of WBC (less than 5 days)
      * At least 10% blasts in blood or marrow
      * At least 20% blasts plus promyelocytes in blood or marrow
      * At least 20% basophils plus eosinophils in blood
      * Anemia or thrombocytopenia unresponsive to busulfan or hydroxyurea
      * Persistent thrombocytosis
      * Additional chromosome changes
      * Increasing splenomegaly
      * Development of chloromas or myelofibrosis
    * Blastic phase

      * At least 30% blasts plus promyelocytes in blood or bone marrow
  * Acute lymphoblastic leukemia
  * Chronic lymphocytic leukemia
  * Myelodysplastic syndromes

    * Refractory anemia with excess blasts (RAEB)
    * Chronic myelomonocytic leukemia
    * RAEB in transformation
  * Multiple myeloma
  * Chronic myeloproliferative diseases including, but not limited to, myelofibrosis with myeloid metaplasia
* Measurable or evaluable disease documented by radiographic, hematologic, bone marrow, or clinical examination parameters
* Refusal of allogeneic bone marrow transplantation allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Albumin at least 2.5 g/dL

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* No other uncontrolled medical disorder
* No active inflammatory bowel disease, ileus, or other chronic malabsorption syndromes
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* At least 3 days since prior hydroxyurea

Endocrine therapy:

* At least 4 weeks since prior systemic steroids for multiple myeloma

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* No prior total gastrectomy or total ileocolectomy

Other:

* No prior tipifarnib
* No concurrent proton pump inhibitors (e.g., omeprazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-08; Primary Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Zimmerman, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Zimmerman TM, Harlin H, Odenike OM, Berk S, Sprague E, Karrison T, Stock W, Larson RA, Ratain MJ, Gajewski TF. Dose-ranging pharmacodynamic study of tipifarnib (R115777) in patients with relapsed and refractory hematologic malignancies. J Clin Oncol. 2004 Dec 1;22(23):4816-22. doi: 10.1200/JCO.2004.03.200. PMID 15570084